CLINICAL TRIAL: NCT01131507
Title: A Multicenter, Open-Label, Safety Extension of Study PR-011 Titled: A Multicenter, Randomized, Open-Label, Crossover Study to Evaluate the Mode of Administration and Safety of EUR-1008 in Infants 1 to 12 Months of Age With Exocrine Pancreatic Insufficiency (EPI) Associated With Cystic Fibrosis (CF)
Brief Title: PR-018: An Open-Label, Safety Extension of Study PR-011
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR-018
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: Exocrine Pancreatic Insufficiency; Infants with CF
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUR-1008 (APT-1008) (Experimental)
  Interventions: Drug: EUR-1008 (APT-1008)

INTERVENTIONS:
Drug: EUR-1008 (APT-1008) — EUR-1008 (APT-1008) (Zenpep® [pancrelipase] 3,000 lipase units delayed release capsules) from open capsules mixed with a small amount of apple juice or apple sauce will be administered orally starting at the same dose as administered at the end of study PR-011 (NCT01100606), with dose increments of 3,000 lipase units. The dose will be adjusted based on participants' age and body weight. Total dose will not exceed 10,000 lipase units per kilogram (kg) of body weight per day unless clinically indicated. Total duration of study treatment will be up to 12 months.
  Other Names: Zenpep® (pancrelipase) 3,000 lipase units delayed release capsules

SUMMARY:
A study to evaluate long term safety and effect on ability to thrive of EUR-1008 (APT-1008) 3,000 lipase units (Zenpep® [pancrelipase] delayed release capsules) in infants with exocrine pancreatic insufficiency (EPI) due to cystic fibrosis (CF).

DETAILED DESCRIPTION:
This is a multi-center, open-label, safety extension of Aptalis (formerly Eurand) study PR-011 (NCT01100606) in pediatric participants with EPI due to CF. The study will be carried out in participants who completed the PR-011 study.

The study is comprised of 5 visits: an enrollment visit, treatment visit 1 (3 months), treatment visit 2 (6 months), treatment visit 3 (9 months) and treatment visit 4 (12 months). Once determined eligible for participation, participants will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant's parent or guardian signed informed consent form (ICF)
* Participants who have completed study PR-011 (NCT01100606)

Exclusion Criteria:

* Participant having any condition that would, in the investigator's opinion, limit the participant's ability to complete the study or will result in excess risk to the participant that is above the standard of care

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aptalis Medical Information, Study Director — Forest Laboratories
Locations (6):
- United States (6):
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Lung Specialists Ltd., Las Vegas, Nevada
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Cystic Fibrosis Care Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed previous study PR-011 (NCT01100606) and consented to continue treatment with EUR-1008 (APT-1008) 3,000 lipase units were enrolled in this study.
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) (Zenpep® [pancrelipase] 3,000 lipase units delayed release capsules) from open capsules mixed with a small amount of apple juice or apple sauce orally starting at the same dose as administered at the end of study PR-011 (NCT01100606), with dose increments of 3,000 lipase units. The dose was adjusted based on participants' age and body weight. Total dose not to exceed 10,000 lipase units per kilogram (kg) of body weight per day unless clinically indicated. Total duration of study treatment was up to 12 months.
Period: Overall Study
Arm/Group | EUR-1008 (APT-1008)
Started | 15
Completed | 12
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least 1 dose of study drug.
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) (Zenpep® [pancrelipase] 3,000 lipase units delayed release capsules) from open capsules mixed with a small amount of apple juice or apple sauce orally starting at the same dose as administered at the end of study PR-011 (NCT01100606), with dose increments of 3,000 lipase units. The dose was adjusted based on participants' age and body weight. Total dose not to exceed 10,000 lipase units per kg body weight per day unless clinically indicated. Total duration of study treatment was up to 12 months.
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: months] | 9.0 (3.27) [3 to 14]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Weight [Median (Full Range); unit: kilogram] | 7.80 (1.296) [6.0 to 10.6]
Length [Median (Full Range); unit: centimeter] — Number of participants evaluable for this baseline characteristic = 14
  centimeter | 68.5 (5.98) [59 to 79]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAE was any event not present prior to exposure to study drug or any event already present that worsened in either intensity or frequency following exposure to test drug. Serious AE (SAE) was any event that resulted in death, immediately life threatening, hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or a congenital anomaly/birth defect. Number of participants with TEAEs, SAEs, TEAE's relationship to study drug (unrelated, possible and probable) and on the basis of severity (mild [minimal/no treatment and did not interfere with daily activities], moderate [resulted in a low level of inconvenience or concern with the therapeutic measures and may have caused some interference with functioning] and severe [interrupted participant's usual daily activity, may have required systemic drug therapy or other treatment and were usually incapacitating]) with a frequency threshold of above 5% were reported.
Time Frame: Up to Month 12 or early termination
Population: Safety population included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 15
participants
  All TEAEs | 15
  SAEs | 3
  Unrelated TEAEs | 10
  Possibly related TEAEs | 4
  Probably related TEAEs | 1
  Mild TEAEs | 5
  Moderate TEAEs | 8
  Severe TEAEs | 2

2. Secondary Outcome: Change From Baseline in Growth Percentiles at Month 3, 6, 9 and 12
Description: Participant's ability to thrive was evaluated through growth percentiles for weight-for-age, length-for-age and weight-for-length recorded on Center for Disease Control and Prevention (CDC) growth charts during each treatment visit.
Time Frame: Baseline, Month 3, 6, 9 and 12
Population: Safety population included all participants who received at least 1 dose of study drug. Here, 'n' specifies number of participants who were evaluable for various categories at each time point.
Measure: Median (Full Range); unit: growth percentile
Arm/Group | EUR-1008 (APT-1008)
Number analyzed (Participants) | 15
growth percentile
  Weight-for-age: Baseline (n=15) | 22.0 [2 to 91]
  Weight-for-age: Change at Month 3 (n=15) | 2.0 [-18 to 34]
  Weight-for-age: Change at Month 6 (n=13) | 6.0 [-35 to 34]
  Weight-for-age: Change at Month 9 (n=12) | 4.0 [-42 to 34]
  Weight-for-age: Change at Month 12 (n=12) | 5.5 [-45 to 36]
  Length-for-age: Baseline (n=14) | 36.5 [1 to 74]
  Length-for-age: Change at Month 3 (n=14) | 2.0 [-22 to 30]
  Length-for-age: Change at Month 6 (n=12) | 2.0 [-23 to 28]
  Length-for-age: Change at Month 9 (n=12) | 11.0 [-24 to 34]
  Length-for-age: Change at Month 12 (n=12) | 0.5 [-27 to 53]
  Weight-for-length: Baseline (n=14) | 41.5 [8 to 98]
  Weight-for-length: Change at Month 3 (n=14) | 0.5 [-12 to 41]
  Weight-for-length: Change at Month 6 (n=12) | 13.5 [-17 to 47]
  Weight-for-length: Change at Month 9 (n=12) | 9.0 [-54 to 31]
  Weight-for-length: Change at Month 12 (n=12) | 10.5 [-57 to 48]

ADVERSE EVENTS:
Time Frame: Up to Month 12 or early termination
Description: Adverse event (AE) was defined as any untoward medical occurrence regardless of causal relationship to study medication. Serious AE was any event that resulted in death, life threatening, required or prolonged in-patient hospitalization, significant disability/incapacity, or was a congenital anomaly/birth defect.
Groups:
- EUR-1008 (APT-1008): EUR-1008 (APT-1008) (Zenpep® [pancrelipase] 3,000 lipase units delayed release capsules) from open capsules mixed with a small amount of apple juice or apple sauce will be administered orally starting at the same dose as administered at the end of study PR-011 (NCT01100606), with dose increments of 3,000 lipase units. The dose was adjusted based on participants' age and body weight. Total dose not to exceed 10,000 lipase units per kg body weight per day unless clinically indicated. Total duration of study treatment was up to 12 months.
Arm/Group | EUR-1008 (APT-1008)
Serious Adverse Events (participants affected / at risk) | 3/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=15)
Bronchopneumonia (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Anaphylactic shock (Immune system disorders) | 1 — This AE was an acute reaction to peanuts and not related to study drug.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EUR-1008 (APT-1008) (N=15)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Steatorrhoea (Gastrointestinal disorders) | 4
Abnormal faeces (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 2
Faecal volume increased (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Post-tussive vomiting (Gastrointestinal disorders) | 2
Teething (Gastrointestinal disorders) | 2
Faeces hard (Gastrointestinal disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Malabsorption (Gastrointestinal disorders) | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Otitis media (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 2
Pseudomonas infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Acute sinusitis (Infections and infestations) | 1
Croup infectious (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Pyrexia (General disorders) | 10
Fatigue (General disorders) | 3
Decreased appetite (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 2
Weight gain poor (Metabolism and nutrition disorders) | 1
Weight decreased (Investigations) | 2
Band neutrophil count increased (Investigations) | 1
Pseudomonas test positive (Investigations) | 1
Cystic fibrosis lung (Congenital, familial and genetic disorders) | 3
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Cerumen impaction (Ear and labyrinth disorders) | 1
Eyelid margin crusting (Eye disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restrictions vary in accordance with each agreement with the individual investigators. Sponsor will allow publication after a multi-center publication has been published or after an agreed period of time if no such multi-center publication is submitted for publication. Sponsor can ask that Sponsor's confidential information be removed from any publication and can defer publication for a period of time to allow for Sponsor to obtain patent or other intellectual property right protection.